CLINICAL TRIAL: NCT06735079
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of REL-1017 As Adjunctive Treatment for Major Depressive Disorder (MDD)
Brief Title: A Study to Evaluate the Efficacy and Safety of REL-1017 As Adjunctive Treatment of Major Depressive Disorder (MDD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn based on business-related matters and there are no new safety concerns related to the trial. No patients were enrolled.
Sponsor: MGGM LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REL-1017-305
Record Dates: First submitted 2024-12-13; First posted 2024-12-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: MDD; Esmethadone; Adjunctive therapy; REL-1017; NMDA
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- REL 1017-305 (Experimental)
  Interventions: Drug: REL1017 (esmethadone HCI) (active drug)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REL1017 (esmethadone HCI) (active drug) — REL-1017 is an investigational drug administered as an oral tablet, once daily. The dosing regimen includes a 75 mg dose on Day 1 (three tablets) in the clinic, followed by 25 mg daily (one tablet) at home from Day 2 to Day 28, with regular safety, efficacy, and tolerability assessments REL-1017 (esmethadone HCl) is under investigation as a novel NMDAR antagonist. Unlike racemic methadone, it lacks opioid-like effects such as dependency or respiratory depression. REL-1017 also lacks dissociative effects seen with more potent NMDAR antagonists such as ketamine. Finally, REL-1017 does not appear to have metabolic or neurological side effects.
  Arms: REL 1017-305
Drug: Placebo — The placebo serves as a control to evaluate the effectiveness and safety of REL-1017. It is an inactive substance that matches the active drug in appearance but contains no active ingredients. The placebo group allows researchers to compare outcomes, such as changes in depressive symptoms, with the active drug group.
  The double-blind design ensures neither participants nor researchers know who is receiving the active treatment or placebo, eliminating bias. The placebo also helps assess whether observed side effects are due to the drug or unrelated factors.
  Participants are randomly assigned to receive either REL-1017 or the placebo, both administered once daily for 28 days. This helps establish REL-1017's clinical effectiveness and safety in treating Major Depressive Disorder (MDD).
  Arms: Placebo

SUMMARY:
Study Overview This clinical trial is a Phase 3 research study designed to test the safety and effectiveness of an investigational drug called REL-1017 (esmethadone HCl). The goal is to determine if REL-1017 can help people with major depressive disorder (MDD) who are already taking other antidepressant medications but have not experienced enough improvement.

Why This Study Is Important MDD is a serious condition that affects mood, cognition, motivation, energy, and daily life. Some people do not respond fully to standard antidepressants. REL-1017 is being tested as an additional treatment to see if it can improve symptoms more effectively.

Who Can Participate The study is enrolling adults diagnosed with major depressive disorder who do not have enough relief from their current antidepressant medications. Specific criteria must be met to join the study.

What Happens in the Study Participants will be randomly assigned to receive either REL-1017 or a placebo (an inactive substance) along with their current antidepressant. This process helps researchers understand the effects of the drug. Neither the participants nor the researchers will know who receives REL-1017 or the placebo during the study.

Study Details Duration: The study involves several weeks of treatment and follow-up visits. Assessments: Participants will complete health evaluations, including physical exams and questionnaires, to monitor progress and side effects.

Costs: Study-related treatments and assessments are provided at no cost to participants.

Potential Benefits and Risks Benefits: Participants may experience improvements in depressive symptoms. Risks: As with any investigational medication, there may be side effects. All participants will be closely monitored by the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female participant, aged 18 to 65 years, inclusive, at Screening.
3. Body mass index (BMI) between 18.5 and 30.0 kg/m2, inclusive, at Screening.
4. Participant understands the study requirements, is willing and able to commit to meet all study requirements, adhere to both approved ADT and study drug regimen, and complete all assessments and all scheduled visits, per Investigator judgment.

Exclusion Criteria:

1. History or presence of clinically significant abnormality as assessed by physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, which in the opinion of the Investigator would jeopardize the safety of the participant or the validity of the study results, including established QT prolongation, long QT syndrome, torsades de pointes, bradyarrhythmia, ventricular tachycardia, uncompensated heart failure (greater than NYHA Class 1 CHF), uncontrolled hypokalemia, or uncontrolled hypomagnesemia.
2. Any medical, psychiatric condition, or social context that, in the opinion of the Investigator, is likely to unfavourably alter the risk-benefit of participant, to interfere with protocol compliance, or to confound safety or efficacy assessments.
3. Triplicate 12-lead ECG with average QTcF ≥450 msec, and/or a QRS interval ≥120 msec at Screening.
4. Poorly controlled diabetes as defined by a glycosylated hemoglobin (HbA1c) >8.5% (69 mmol/mol), despite standard care. (Note: re-screening of patients who has failed the screening process due to not meeting this exclusion criterion is allowed after diabetes treatment adjustment and level of glycosylated hemoglobin (HbA1c) back to <8.5%)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-27 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
MADRS10 | 28 days
  To evaluate the therapeutic efficacy of REL-1017 compared to placebo in participants with inadequate response to ongoing ADT at Day 28 on the Montgomery-Åsberg Depression Rating Scale (MADRS10) total score.
  Scale: Montgomery-Åsberg Depression Rating Scale (MADRS)
  Minimum and Maximum Values: The scale ranges from 0 to 60. Interpretation of Higher Scores: Higher scores indicate greater severity of depression.
  Specific Ranges:
  0-6: Normal/no symptoms. 7-19: Mild depression. 20-34: Moderate depression. 35-60: Severe depression.

SECONDARY OUTCOMES:
MADRS10 | 7 days
  Decrease from Baseline to Day 7 of the MADRS10 total score
  Scale: Montgomery-Åsberg Depression Rating Scale (MADRS)
MADRS10 | 28 days
  MADRS10 response rate (improvement ≥50% compared with total Baseline score) at Day 28
  Scale: Montgomery-Åsberg Depression Rating Scale (MADRS)
MADRS10 | 28 days
  MADRS10 remission rate (total score ≤10) at Day 28
  Scale: Montgomery-Åsberg Depression Rating Scale (MADRS)
CGI-S | 28 days
  Decrease from Baseline to Day 28 of the CGI-S score
  Scale: CGI-S
  The CGI-S measures the severity of the disease using a 7-point Likert scale ranging from 1=normal, not at all ill to 7=among the most extremely ill participants

CONTACTS AND LOCATIONS:
Locations (2):
- Mediolanum Cardio Research, Milan, Italy, Italy
- Clinical Trial Unit - Ente Ospedaliero Cantonale (CTU-EOC) Area Formazione medica e Ricerca (AFRi), Lugano, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: No